CLINICAL TRIAL: NCT03015220
Title: Safety and Efficacy of Oral Semaglutide Versus Dulaglutide Both in Combination With One OAD in Japanese Subjects With Type 2 Diabetes
Brief Title: Safety and Efficacy of Oral Semaglutide Versus Dulaglutide Both in Combination With One OAD (Oral Antidiabetic Drug) in Japanese Subjects With Type 2 Diabetes
Acronym: PIONEER 10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4282; U1111-1181-4133 (Other: WHO); JapicCTI-173485 (Other: Japic)
Record Dates: First submitted 2017-01-06; First posted 2017-01-09 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral semaglutide 3 mg (Experimental)
  Interventions: Drug: Semaglutide
- Oral semaglutide 7 mg (Experimental)
  Interventions: Drug: Semaglutide
- Oral semaglutide 14 mg (Experimental)
  Interventions: Drug: Semaglutide
- Dulaglutide 0.75 mg (Active Comparator)
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Semaglutide — Oral administration once-daily, as add-on to pre-trial oral antidiabetic drug (OAD).
  Arms: Oral semaglutide 14 mg; Oral semaglutide 3 mg; Oral semaglutide 7 mg
Drug: Dulaglutide — Subcutaneously administration (s.c., under the skin) once-weekly, as add-on to pre-trial oral antidiabetic drug (OAD).
  Arms: Dulaglutide 0.75 mg

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate Safety and efficacy of oral semaglutide versus dulaglutide both in combination with one OAD (oral antidiabetic drug) in Japanese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Japanese male or female, age above or equal to 20 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus for at least 60 days prior to day of screening
* HbA1c (glycosylated haemoglobin) between 7.0%-10.5% (53-91 mmol/mol) (both inclusive)
* OAD (oral antidiabetic drug) monotherapy with stable daily dose for at least 60 days prior to the day of screening of one of SU (sulphonylurea) glinide , TZD (thiazolidinedione), α-GI (alpha-glucosidase inhibitor) or SGLT-2 (sodium-glucose cotransporter-2) inhibitor according to Japanese labelling

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method. Adequate contraceptive measures are abstinence (not having sex), diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of multiple endocrine neoplasia type 2 (MEN 2) or medullary thyroid carcinoma (MTC)
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack (TIA) within the past 180 days prior to the day of screening and randomisation
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with alanine aminotransferase (ALT) above 2.5 x upper normal limit (UNL)
* Renal impairment defined as estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)
* Treatment with once-weekly glucagon-like peptide-1 receptor agonists (GLP-1 RA) or once weekly dipeptidyl peptidase-4 (DPP-4) inhibitor in a period of 90 days before the day of screening
* For subjects treated with an OAD other than TZD at screening: Treatment with TZD in a period of 90 days before the day of screening
* Treatment with any medication for the indication of diabetes or obesity in addition to background OAD medication (SU, glinide, TZD, α-GI or SGLT-2 inhibitor) in a period of 60 days before the day of screening with the exception of short-term insulin treatment for acute illness for a total of at least 14 days
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in situ carcinomas)
* History of diabetic ketoacidosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- Japan (31):
  - Novo Nordisk Investigational Site, Adachi-ku, Tokyo
  - Novo Nordisk Investigational Site, Annaka-shi, Gunma
  - Novo Nordisk Investigational Site, Arakawa-ku, Tokyo
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Gunma
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kawaguchi-shi, Saitama
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Kurashiki-shi, Okayama
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Mitaka-shi, Tokyo
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Sapporo
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinagawa-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Toshima-ku, Tokyo
  - Novo Nordisk Investigational Site, Yamato-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitent on novonordisk-trials.com
URL: http://novonordisk-trials.com/

REFERENCES:
- [Result] Ishii H, Hansen BB, Langer J, Horio H. Effect of Orally Administered Semaglutide Versus Dulaglutide on Diabetes-Related Quality of Life in Japanese Patients with Type 2 Diabetes: The PIONEER 10 Randomized, Active-Controlled Trial. Diabetes Ther. 2021 Feb;12(2):613-623. doi: 10.1007/s13300-020-00985-w. Epub 2021 Jan 18. PMID 33460016
- [Result] Yabe D, Nakamura J, Kaneto H, Deenadayalan S, Navarria A, Gislum M, Inagaki N; PIONEER 10 Investigators. Safety and efficacy of oral semaglutide versus dulaglutide in Japanese patients with type 2 diabetes (PIONEER 10): an open-label, randomised, active-controlled, phase 3a trial. Lancet Diabetes Endocrinol. 2020 May;8(5):392-406. doi: 10.1016/S2213-8587(20)30074-7. PMID 32333876
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 36 sites in Japan.
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Participants were to take oral semaglutide 3 mg tablets once-daily from week 0 to week 52. In addition, participants were to continue their pre-trial oral anti-diabetic drug (OAD) (either of sulphonylurea, glinide, thiazolidinedione, alpha-glucosidase inhibitor or SGLT-2 inhibitor) from week 0 to week 52.
- Oral Semaglutide 7 mg: Participants were to take oral semaglutide tablets once-daily in a dose escalation manner from week 0 to week 52: 3 mg from week 0 to week 4 and 7 mg from week 4 to week 52. In addition, participants were to continue their pre-trial OAD (either of sulphonylurea, glinide, thiazolidinedione, alpha-glucosidase inhibitor or SGLT-2 inhibitor) from week 0 to week 52.
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once-daily in a dose escalation manner from week 0 to week 52: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 52. In addition, participants were to continue their pre-trial OAD (either of sulphonylurea, glinide, thiazolidinedione, alpha-glucosidase inhibitor or SGLT-2 inhibitor) from week 0 to week 52.
- Dulaglutide 0.75 mg: Participants were to take dulaglutide 0.75 mg subcutaneous (under the skin) injections once-weekly from week 0 to week 52. In addition, participants were to continue their pre-trial OAD (either of sulphonylurea, glinide, thiazolidinedione, alpha-glucosidase inhibitor or SGLT-2 inhibitor) from week 0 to week 52.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Started | 131 | 132 | 130 | 65
Full Analysis Set (FAS) | 131 | 132 | 130 | 65
Safety Analysis Set (SAS) | 131 | 132 | 130 | 65
Completed | 128 | 130 | 127 | 63
Not Completed | 3 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The FAS comprised of all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg | Total
Number analyzed (Participants) | 131 | 132 | 130 | 65 | 458
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (10) | 58 (11) | 57 (10) | 61 (9) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 42 | 30 | 14 | 117
  Male | 100 | 90 | 100 | 51 | 341
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 131 | 132 | 130 | 65 | 458
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 131 | 132 | 130 | 65 | 458
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 57 (52-week treatment period plus the 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Events | 330 | 350 | 324 | 178

2. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Percentage of HbA1c
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | -1.1 (0.9) | -1.7 (0.9) | -2.0 (1.0) | -1.6 (0.9)
  Week 52: number analyzed (Participants) | 126 | 129 | 127 | 63
  Week 52 | -0.8 (1.0) | -1.4 (1.0) | -1.8 (1.0) | -1.4 (0.9)

3. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
mmol/L
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | -1.23 (1.54) | -2.25 (1.93) | -2.72 (1.86) | -2.22 (1.71)
  Week 52: number analyzed (Participants) | 125 | 128 | 127 | 63
  Week 52 | -0.95 (1.72) | -1.96 (1.72) | -2.18 (2.50) | -1.80 (1.71)

4. Secondary Outcome: Change in Self-measured Plasma Glucose 7-point Profile (SMPG) - Mean 7-point Profile
Description: Change from baseline (week 0) in mean 7-point SMPG profile was evaluated at weeks 26 and 52. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
mmol/L
  Week 26: number analyzed (Participants) | 126 | 128 | 127 | 64
  Week 26 | -1.8 (2.2) | -2.7 (2.1) | -3.5 (2.3) | -2.9 (2.4)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 62
  Week 52 | -1.7 (2.1) | -2.5 (2.4) | -3.3 (2.6) | -2.6 (2.6)

5. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG) - Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) in the average of the post-prandial increments over all meals was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
mmol/L
  Week 26: number analyzed (Participants) | 127 | 128 | 127 | 64
  Week 26 | -0.9 (2.5) | -1.3 (2.0) | -1.2 (2.4) | -0.7 (2.3)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 62
  Week 52 | -0.6 (2.6) | -0.8 (2.0) | -0.9 (2.6) | -0.7 (2.3)

6. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
kg
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | -0.1 (2.0) | -1.0 (3.0) | -2.2 (3.2) | 0.3 (2.1)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52 | 0.0 (2.4) | -0.9 (3.4) | -1.7 (3.5) | 1.0 (2.7)

7. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Percentage change
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | -0.28 (2.79) | -1.49 (4.25) | -3.21 (4.32) | 0.25 (3.33)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52 | -0.02 (3.28) | -1.34 (4.77) | -2.33 (4.67) | 1.25 (4.06)

8. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline (week 0) in BMI was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Kilogram per square meter (kg/m^2)
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | -0.1 (0.7) | -0.4 (1.1) | -0.8 (1.2) | 0.1 (0.8)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52 | -0.0 (0.9) | -0.3 (1.3) | -0.6 (1.3) | 0.3 (1.0)

9. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at weeks 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Centimeters (cm)
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26 | 0.0 (3.1) | -0.6 (3.4) | -1.2 (4.3) | 0.3 (2.9)
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52 | -0.1 (3.6) | -0.8 (3.9) | -1.7 (4.2) | 0.7 (3.6)

10. Secondary Outcome: Change in Fasting Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting total cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of fasting total cholesterol
  Week 26: number analyzed (Participants) | 126 | 127 | 128 | 63
  Week 26 | 0.96 (9.4) | 0.91 (12.3) | 0.91 (12.3) | 0.92 (8.8)
  Week 52: number analyzed (Participants) | 124 | 127 | 126 | 62
  Week 52 | 0.98 (12.7) | 0.95 (13.3) | 0.94 (12.5) | 0.93 (11.4)

11. Secondary Outcome: Change in Fasting Low-density Lipoprotein (LDL) - Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting low-density lipoprotein (LDL) (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting LDL
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of fasting LDL
  Week 26: number analyzed (Participants) | 126 | 127 | 128 | 63
  Week 26 | 0.92 (15.9) | 0.88 (18.4) | 0.87 (20.7) | 0.88 (14.5)
  Week 52: number analyzed (Participants) | 124 | 127 | 126 | 62
  Week 52 | 0.98 (17.4) | 0.94 (19.0) | 0.92 (18.6) | 0.91 (16.2)

12. Secondary Outcome: Change in Fasting High-density Lipoprotein (HDL) - Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting high-density lipoprotein (HDL) (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting HDL
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of fasting HDL
  Week 26: number analyzed (Participants) | 126 | 127 | 128 | 63
  Week 26 | 1.02 (13.1) | 0.99 (12.8) | 1.00 (12.5) | 0.99 (11.6)
  Week 52: number analyzed (Participants) | 124 | 127 | 126 | 62
  Week 52 | 1.03 (11.2) | 0.99 (14.5) | 1.01 (13.1) | 1.00 (11.6)

13. Secondary Outcome: Change in Fasting Very-low Density Lipoprotein (VLDL) - Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting very-low density lipoprotein (VLDL) (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting VLDL
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of fasting VLDL
  Week 26: number analyzed (Participants) | 126 | 127 | 128 | 63
  Week 26 | 1.03 (37.9) | 0.92 (32.3) | 0.96 (33.6) | 0.93 (33.5)
  Week 52: number analyzed (Participants) | 124 | 127 | 126 | 62
  Week 52 | 0.90 (33.3) | 0.87 (39.4) | 0.86 (36.9) | 0.88 (31.6)

14. Secondary Outcome: Change in Fasting Triglyceride (Ratio to Baseline)
Description: Change from baseline (week 0) in fasting triglycerides (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of fasting triglycerides
  Week 26: number analyzed (Participants) | 126 | 127 | 128 | 63
  Week 26 | 1.03 (41.1) | 0.91 (34.1) | 0.96 (34.0) | 0.93 (33.7)
  Week 52: number analyzed (Participants) | 124 | 127 | 126 | 62
  Week 52 | 0.89 (33.9) | 0.87 (43.0) | 0.87 (38.3) | 0.88 (30.8)

15. Secondary Outcome: Participants Who Achieve HbA1c Below 7% (53 mmol/Mol), American Diabetes Association Target (Yes/No)
Description: Participants who achieved HbA1c below 7.0% (53 millimoles per mole [mmol/mol]) according to American Diabetes Association (ADA) target (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 59 | 96 | 105 | 45
  Week 26: No | 69 | 32 | 23 | 19
  Week 52: number analyzed (Participants) | 126 | 129 | 127 | 63
  Week 52: Yes | 43 | 77 | 90 | 32
  Week 52: No | 83 | 52 | 37 | 31

16. Secondary Outcome: Participants Who Achieve HbA1c Below or Equal to 6.5% (48 mmol/Mol), American Association of Clinical Endocrinologists Target (Yes/No)
Description: Participants who achieved HbA1c below or equal to 6.5% (48 mmol/mol), American Association of Clinical Endocrinologists (AACE) target (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 40 | 67 | 88 | 31
  Week 26: No | 88 | 61 | 40 | 33
  Week 52: number analyzed (Participants) | 126 | 129 | 127 | 63
  Week 52: Yes | 22 | 50 | 69 | 23
  Week 52: No | 104 | 79 | 58 | 40

17. Secondary Outcome: Participants Who Achieve HbA1c Below 7.0% (53 mmol/Mol) Without Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain (Yes/No)
Description: Participants who achieved HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia episodes and without weight gain (yes/no) at weeks 26 and 52 are presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 39 | 63 | 84 | 25
  Week 26: No | 89 | 65 | 44 | 39
  Week 52: number analyzed (Participants) | 126 | 129 | 127 | 63
  Week 52: Yes | 23 | 53 | 71 | 16
  Week 52: No | 103 | 76 | 56 | 47

18. Secondary Outcome: Participants Who Achieve HbA1c Reduction More Than or Equal to 1% (10.9 mmol/Mol) and Weight Loss More Than or Equal to 3% (Yes/No)
Description: Participants who achieved HbA1c reduction more than or equal to 1% (10.9 mmol/mol) and weight loss more than or equal to 3% (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 15 | 34 | 62 | 8
  Week 26: No | 113 | 94 | 66 | 56
  Week 52: number analyzed (Participants) | 126 | 129 | 127 | 63
  Week 52: Yes | 11 | 32 | 42 | 7
  Week 52: No | 115 | 97 | 85 | 56

19. Secondary Outcome: Participants Who Achieve Weight Loss More Than or Equal to 5% (Yes/No).
Description: Participants who achieved weight loss more than or equal to 5% (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 6 | 23 | 39 | 4
  Week 26: No | 122 | 105 | 89 | 60
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52: Yes | 7 | 21 | 28 | 4
  Week 52: No | 120 | 108 | 99 | 59

20. Secondary Outcome: Participants Who Achieve Weight Loss More Than or Equal to 10% (Yes/No)
Description: Participants who achieved weight loss more than or equal to 10% (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 26: number analyzed (Participants) | 128 | 128 | 128 | 64
  Week 26: Yes | 0 | 6 | 8 | 1
  Week 26: No | 128 | 122 | 120 | 63
  Week 52: number analyzed (Participants) | 127 | 129 | 127 | 63
  Week 52: Yes | 0 | 9 | 7 | 0
  Week 52: No | 127 | 120 | 120 | 63

21. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 0 to week 26 | 1 | 3 | 6 | 1
  Week 0 to week 52 | 24 | 13 | 8 | 8
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Dulaglutide 0.75 mg; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment and strata as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.2963, Regression, Cox — Unadjusted two-sided p-value for the test of no difference from 1; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [0.70 to 3.20] — Oral Semaglutide 3 mg /Dulaglutide 0.75 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Dulaglutide 0.75 mg; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.5997, Regression, Cox — Unadjusted two-sided p-value for the test of no difference from 1; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.35 to 1.83] — Oral Semaglutide 7 mg /Dulaglutide 0.75 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Dulaglutide 0.75 mg; [analysis description as in outcome 21, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1871, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.23 to 1.33] — Oral Semaglutide 14 mg /Dulaglutide 0.75 mg

22. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Week 0 to week 26 | 0 | 0 | 1 | 1
  Week 0 to week 52 | 22 | 8 | 2 | 6
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Dulaglutide 0.75 mg; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment and strata as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1672, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 1.90, 95% CI 2-sided [0.76 to 4.72] — Oral Semaglutide 3 mg /Dulaglutide 0.75 mg
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Dulaglutide 0.75 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.3391, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.21 to 1.72] — Oral Semaglutide 7 mg /Dulaglutide 0.75 mg
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Dulaglutide 0.75 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0110, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.12, 95% CI 2-sided [0.02 to 0.62] — Oral Semaglutide 14 mg /Dulaglutide 0.75 mg

23. Secondary Outcome: Change in Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in amylase (measured as units per liter [U/L]) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of amylase
  Week 26: number analyzed (Participants) | 125 | 123 | 121 | 62
  Week 26 | 1.01 (15.1) | 1.07 (18.1) | 1.10 (19.4) | 1.05 (23.4)
  Week 52: number analyzed (Participants) | 123 | 122 | 113 | 60
  Week 52 | 1.03 (18.5) | 1.10 (23.8) | 1.11 (20.0) | 1.07 (18.8)

24. Secondary Outcome: Change in Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (measured as U/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Ratio of lipase
  Week 26: number analyzed (Participants) | 125 | 123 | 121 | 62
  Week 26 | 1.15 (37.4) | 1.27 (35.8) | 1.40 (42.8) | 1.14 (48.3)
  Week 52: number analyzed (Participants) | 123 | 122 | 113 | 60
  Week 52 | 1.11 (34.7) | 1.36 (50.3) | 1.40 (42.0) | 1.15 (57.7)

25. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at weeks 26 and 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Beats per minute (beats/min)
  Week 26: number analyzed (Participants) | 126 | 124 | 121 | 63
  Week 26 | 3 (9) | 4 (10) | 4 (9) | 4 (9)
  Week 52: number analyzed (Participants) | 124 | 123 | 114 | 61
  Week 52 | 3 (10) | 3 (9) | 3 (9) | 2 (10)

26. Secondary Outcome: Change in Blood Pressure
Description: Change from baseline (week 0) in blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) was evaluated at weeks 26 and 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Millimeters of mercury (mmHg)
  Week 26: SBP: number analyzed (Participants) | 126 | 124 | 121 | 63
  Week 26: SBP | -3.0 (13.0) | -5.0 (13.0) | -6.0 (15.0) | -4.0 (12.0)
  Week 52: SBP: number analyzed (Participants) | 124 | 123 | 114 | 61
  Week 52: SBP | -2.0 (14.0) | -2.0 (13.0) | -2.0 (13.0) | -3.0 (13.0)
  Week 26: DBP: number analyzed (Participants) | 126 | 124 | 121 | 63
  Week 26: DBP | -1.0 (9.0) | -1.0 (9.0) | -2.0 (10.0) | -1.0 (11.0)
  Week 52: DBP | 0.0 (9.0) | 0.0 (9.0) | -1.0 (10.0) | 0.0 (9.0)

27. Secondary Outcome: Change in ECG Evaluation
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at weeks 26 and 52. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS) and abnormal and clinically significant (CS)) from week 0 to week 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 109 | 113 | 102 | 58
  Normal (week 0) to normal (week 26) | 103 | 110 | 99 | 54
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 109 | 113 | 102 | 58
  Normal (week 0) to abnormal NCS (week 26) | 4 | 3 | 3 | 4
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 109 | 113 | 102 | 58
  Normal (week 0) to abnormal CS (week 26) | 2 | 0 | 0 | 0
  Abnormal NCS (week 0) to normal (week 26): number analyzed (Participants) | 16 | 15 | 24 | 6
  Abnormal NCS (week 0) to normal (week 26) | 0 | 3 | 4 | 2
  Abnormal NCS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 16 | 15 | 24 | 6
  Abnormal NCS (week 0) to abnormal NCS (week 26) | 16 | 12 | 18 | 4
  Abnormal NCS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 16 | 15 | 24 | 6
  Abnormal NCS (week 0) to abnormal CS (week 26) | 0 | 0 | 2 | 0
  Abnormal CS (week 0) to normal (week 26): number analyzed (Participants) | 3 | 1 | 2 | 0
  Abnormal CS (week 0) to normal (week 26) | 1 | 0 | 0 | 0
  Abnormal CS (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 3 | 1 | 2 | 0
  Abnormal CS (week 0) to abnormal NCS (week 26) | 0 | 0 | 0 | 0
  Abnormal CS (week 0) to abnormal CS (week 26): number analyzed (Participants) | 3 | 1 | 2 | 0
  Abnormal CS (week 0) to abnormal CS (week 26) | 2 | 1 | 2 | 0
  Normal (week 0) to normal (week 52): number analyzed (Participants) | 108 | 113 | 102 | 57
  Normal (week 0) to normal (week 52) | 103 | 108 | 95 | 55
  Normal (week 0) to abnormal NCS (week 52): number analyzed (Participants) | 108 | 113 | 102 | 57
  Normal (week 0) to abnormal NCS (week 52) | 3 | 5 | 6 | 2
  Normal (week 0) to abnormal CS (week 52): number analyzed (Participants) | 108 | 113 | 102 | 57
  Normal (week 0) to abnormal CS (week 52) | 2 | 0 | 1 | 0
  Abnormal (week 0) NCS to normal (week 52): number analyzed (Participants) | 15 | 15 | 24 | 6
  Abnormal (week 0) NCS to normal (week 52) | 2 | 5 | 6 | 3
  Abnormal (week 0) NCS to abnormal NCS (week 52): number analyzed (Participants) | 15 | 15 | 24 | 6
  Abnormal (week 0) NCS to abnormal NCS (week 52) | 13 | 10 | 18 | 3
  Abnormal (week 0) NCS to abnormal CS (week 52): number analyzed (Participants) | 15 | 15 | 24 | 6
  Abnormal (week 0) NCS to abnormal CS (week 52) | 0 | 0 | 0 | 0
  Abnormal (week 0) CS to normal (week 52): number analyzed (Participants) | 4 | 1 | 1 | 0
  Abnormal (week 0) CS to normal (week 52) | 1 | 1 | 0 | 0
  Abnormal (week 0) CS to abnormal NCS (week 52): number analyzed (Participants) | 4 | 1 | 1 | 0
  Abnormal (week 0) CS to abnormal NCS (week 52) | 0 | 0 | 0 | 0
  Abnormal (week 0) CS to abnormal CS (week 52): number analyzed (Participants) | 4 | 1 | 1 | 0
  Abnormal (week 0) CS to abnormal CS (week 52) | 3 | 0 | 1 | 0

28. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (weeks -2), week 26 and weeks 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Central and peripheral nervous system; 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head, ears, eyes, nose, throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week -2, week 26, week 52
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  1) Cardiovascular system (week -2): Normal | 128 | 132 | 128 | 60
  1) Cardiovascular system (week -2): Abnormal NCS | 1 | 0 | 0 | 1
  1) Cardiovascular system (week -2): Abnormal CS | 2 | 0 | 2 | 4
  1) Cardiovascular system (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  1) Cardiovascular system (week 26): Normal | 125 | 128 | 125 | 59
  1) Cardiovascular system (week 26): Abnormal NCS | 0 | 0 | 1 | 1
  1) Cardiovascular system (week 26): Abnormal CS | 3 | 0 | 2 | 4
  1) Cardiovascular system (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  1) Cardiovascular system (week 52): Normal | 124 | 129 | 126 | 58
  1) Cardiovascular system (week 52): Abnormal NCS | 1 | 0 | 0 | 1
  1) Cardiovascular system (week 52): Abnormal CS | 2 | 0 | 1 | 4
  2) Central and peripheral nervous system (week -2): Normal | 131 | 131 | 130 | 64
  2) Central and peripheral nervous system (week -2): Abnormal NCS | 0 | 1 | 0 | 0
  2) Central and peripheral nervous system (week -2): Abnormal CS | 0 | 0 | 0 | 1
  2) Central and peripheral nervous system (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  2) Central and peripheral nervous system (week 26): Normal | 128 | 127 | 128 | 62
  2) Central and peripheral nervous system (week 26): Abnormal NCS | 0 | 0 | 0 | 0
  2) Central and peripheral nervous system (week 26): Abnormal CS | 0 | 1 | 0 | 2
  2) Central and peripheral nervous system (week 56): number analyzed (Participants) | 127 | 129 | 127 | 63
  2) Central and peripheral nervous system (week 56): Normal | 127 | 128 | 126 | 62
  2) Central and peripheral nervous system (week 56): Abnormal NCS | 0 | 0 | 0 | 0
  2) Central and peripheral nervous system (week 56): Abnormal CS | 0 | 1 | 1 | 1
  3) Gastrointestinal system, incl. mouth (week -2): Normal | 126 | 128 | 129 | 60
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal NCS | 0 | 2 | 0 | 0
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal CS | 5 | 2 | 1 | 5
  3) Gastrointestinal system, incl. mouth (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  3) Gastrointestinal system, incl. mouth (week 26): Normal | 122 | 123 | 125 | 60
  3) Gastrointestinal system, incl. mouth (week 26): Abnormal NCS | 0 | 2 | 1 | 0
  3) Gastrointestinal system, incl. mouth (week 26): Abnormal CS | 6 | 3 | 2 | 4
  3) Gastrointestinal system, incl. mouth (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  3) Gastrointestinal system, incl. mouth (week 52): Normal | 122 | 124 | 126 | 59
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal NCS | 1 | 3 | 1 | 0
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal CS | 4 | 2 | 0 | 4
  4.General appearance (week -2): Normal | 131 | 132 | 130 | 64
  4.General appearance (week -2): Abnormal NCS | 0 | 0 | 0 | 1
  4.General appearance (week -2): Abnormal CS | 0 | 0 | 0 | 0
  4.General appearance (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  4.General appearance (week 26): Normal | 127 | 128 | 127 | 62
  4.General appearance (week 26): Abnormal NCS | 1 | 0 | 1 | 1
  4.General appearance (week 26): Abnormal CS | 0 | 0 | 0 | 1
  4.General appearance (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  4.General appearance (week 52): Normal | 126 | 128 | 127 | 62
  4.General appearance (week 52): Abnormal NCS | 0 | 0 | 0 | 1
  4.General appearance (week 52): Abnormal CS | 1 | 1 | 0 | 0
  5.Head, ears, eyes, nose, throat, neck (week -2): Normal | 121 | 127 | 124 | 55
  5.Head, ears, eyes, nose, throat, neck (week -2): Abnormal NCS | 3 | 2 | 2 | 4
  5.Head, ears, eyes, nose, throat, neck (week -2): Abnormal CS | 7 | 3 | 4 | 6
  5.Head, ears, eyes, nose, throat, neck (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  5.Head, ears, eyes, nose, throat, neck (week 26): Normal | 119 | 122 | 125 | 56
  5.Head, ears, eyes, nose, throat, neck (week 26): Abnormal NCS | 4 | 1 | 1 | 3
  5.Head, ears, eyes, nose, throat, neck (week 26): Abnormal CS | 5 | 5 | 2 | 5
  5.Head, ears, eyes, nose, throat, neck (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  5.Head, ears, eyes, nose, throat, neck (week 52): Normal | 117 | 123 | 122 | 53
  5.Head, ears, eyes, nose, throat, neck (week 52): Abnormal NCS | 3 | 1 | 2 | 4
  5.Head, ears, eyes, nose, throat, neck (week 52): Abnormal CS | 7 | 5 | 3 | 6
  6. Lymph node palpation (week -2): Normal | 131 | 131 | 129 | 65
  6. Lymph node palpation (week -2): Abnormal NCS | 0 | 1 | 1 | 0
  6. Lymph node palpation (week -2): Abnormal CS | 0 | 0 | 0 | 0
  6. Lymph node palpation (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  6. Lymph node palpation (week 26): Normal | 128 | 127 | 128 | 64
  6. Lymph node palpation (week 26): Abnormal NCS | 0 | 0 | 0 | 0
  6. Lymph node palpation (week 26): Abnormal CS | 0 | 1 | 0 | 0
  6. Lymph node palpation (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  6. Lymph node palpation (week 52): Normal | 127 | 128 | 127 | 63
  6. Lymph node palpation (week 52): Abnormal NCS | 0 | 1 | 0 | 0
  6. Lymph node palpation (week 52): Abnormal CS | 0 | 0 | 0 | 0
  7. Musculoskeletal system (week -2): Normal | 128 | 126 | 127 | 64
  7. Musculoskeletal system (week -2): Abnormal NCS | 1 | 3 | 2 | 0
  7. Musculoskeletal system (week -2): Abnormal CS | 2 | 3 | 1 | 1
  7. Musculoskeletal system (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  7. Musculoskeletal system (week 26): Normal | 123 | 123 | 124 | 61
  7. Musculoskeletal system (week 26): Abnormal NCS | 2 | 2 | 2 | 0
  7. Musculoskeletal system (week 26): Abnormal CS | 3 | 3 | 2 | 3
  7. Musculoskeletal system (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  7. Musculoskeletal system (week 52): Normal | 120 | 125 | 123 | 62
  7. Musculoskeletal system (week 52): Abnormal NCS | 4 | 1 | 2 | 0
  7. Musculoskeletal system (week 52): Abnormal CS | 3 | 3 | 2 | 1
  8) Respiratory system (week -2): Normal | 131 | 132 | 130 | 64
  8) Respiratory system (week -2): Abnormal NCS | 0 | 0 | 0 | 0
  8) Respiratory system (week -2): Abnormal CS | 0 | 0 | 0 | 1
  8) Respiratory system (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  8) Respiratory system (week 26): Normal | 128 | 127 | 128 | 62
  8) Respiratory system (week 26): Abnormal NCS | 0 | 0 | 0 | 0
  8) Respiratory system (week 26): Abnormal CS | 0 | 1 | 0 | 2
  8) Respiratory system (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  8) Respiratory system (week 52): Normal | 126 | 127 | 127 | 62
  8) Respiratory system (week 52): Abnormal NCS | 0 | 1 | 0 | 0
  8) Respiratory system (week 52): Abnormal CS | 1 | 1 | 0 | 1
  9) Skin (week -2): Normal | 125 | 127 | 128 | 63
  9) Skin (week -2): Abnormal NCS | 3 | 0 | 1 | 0
  9) Skin (week -2): Abnormal CS | 3 | 5 | 1 | 2
  9) Skin (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  9) Skin (week 26): Normal | 124 | 127 | 126 | 62
  9) Skin (week 26): Abnormal NCS | 1 | 0 | 1 | 1
  9) Skin (week 26): Abnormal CS | 3 | 1 | 1 | 1
  9) Skin (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  9) Skin (week 52): Normal | 123 | 127 | 125 | 61
  9) Skin (week 52): Abnormal NCS | 1 | 1 | 1 | 0
  9) Skin (week 52): Abnormal CS | 3 | 1 | 1 | 2
  10) Thyroid gland (week -2): Normal | 130 | 130 | 129 | 64
  10) Thyroid gland (week -2): Abnormal NCS | 0 | 2 | 0 | 0
  10) Thyroid gland (week -2): Abnormal CS | 1 | 0 | 1 | 1
  10) Thyroid gland (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  10) Thyroid gland (week 26): Normal | 128 | 128 | 128 | 63
  10) Thyroid gland (week 26): Abnormal NCS | 0 | 0 | 0 | 0
  10) Thyroid gland (week 26): Abnormal CS | 0 | 0 | 0 | 1
  10) Thyroid gland (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  10) Thyroid gland (week 52): Normal | 127 | 129 | 127 | 62
  10) Thyroid gland (week 52): Abnormal NCS | 0 | 0 | 0 | 0
  10) Thyroid gland (week 52): Abnormal CS | 0 | 0 | 0 | 1

29. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination (fundoscopy) findings, normal, abnormal NCS and abnormal CS at baseline (week -2) and week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week -2, week 52
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants
  Left eye (week -2): Normal | 96 | 97 | 90 | 48
  Left eye (week -2): Abnormal NCS | 7 | 2 | 2 | 4
  Left eye (week -2): Abnormal CS | 28 | 33 | 38 | 13
  Left eye (week 52): number analyzed (Participants) | 126 | 129 | 127 | 63
  Left eye (week 52): Normal | 90 | 92 | 93 | 46
  Left eye (week 52): Abnormal NCS | 10 | 8 | 3 | 3
  Left eye (week 52): Abnormal CS | 26 | 29 | 31 | 14
  Right eye (week -2): Normal | 94 | 98 | 89 | 44
  Right eye (week -2): Abnormal NCS | 6 | 3 | 2 | 6
  Right eye (week -2): Abnormal CS | 31 | 31 | 39 | 15
  Right eye (week 52): number analyzed (Participants) | 126 | 129 | 127 | 63
  Right eye (week 52): Normal | 93 | 90 | 90 | 48
  Right eye (week 52): Abnormal NCS | 9 | 8 | 6 | 4
  Right eye (week 52): Abnormal CS | 24 | 31 | 31 | 11

30. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-57 (52-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Episodes | 4 | 4 | 4 | 0

31. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Participants with treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded from week 0 to week 83 (78-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-57
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Participants | 3 | 3 | 4 | 0

32. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey Scores: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at weeks 26 and 52. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Score on a scale
  1) Physical functioning (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  1) Physical functioning (week 26) | -0.18 (3.34) | 0.08 (4.04) | -0.06 (4.16) | -0.24 (3.71)
  1) Physical functioning (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  1) Physical functioning (week 52) | -0.37 (3.34) | 0.70 (4.08) | -0.02 (4.27) | -0.61 (5.01)
  2) Role Physical (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  2) Role Physical (week 26) | -0.58 (5.12) | 0.59 (5.49) | -1.01 (6.00) | -0.48 (5.22)
  2) Role Physical (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  2) Role Physical (week 52) | -0.92 (5.66) | 0.05 (6.13) | -0.92 (7.26) | -0.28 (5.31)
  3) Bodily Pain (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  3) Bodily Pain (week 26) | -0.88 (8.39) | 0.05 (8.26) | -0.99 (9.32) | -0.44 (7.25)
  3) Bodily Pain (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  3) Bodily Pain (week 52) | -2.72 (9.74) | -0.27 (8.88) | 0.01 (9.48) | 0.24 (5.77)
  4)General Health (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  4)General Health (week 26) | 0.42 (4.59) | 0.09 (5.26) | 0.71 (5.94) | -1.03 (5.28)
  4)General Health (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  4)General Health (week 52) | -0.34 (5.27) | 0.01 (5.27) | 0.59 (6.13) | -0.97 (6.63)
  5) Vitality (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  5) Vitality (week 26) | -1.62 (7.49) | -0.79 (7.08) | -0.83 (6.84) | -1.40 (7.94)
  5) Vitality (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  5) Vitality (week 52) | -0.90 (7.29) | -0.11 (7.03) | 0.09 (6.83) | -0.86 (7.63)
  6) Social functioning (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  6) Social functioning (week 26) | -0.77 (5.87) | -0.15 (5.95) | -0.15 (6.08) | 0.15 (4.98)
  6) Social functioning (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  6) Social functioning (week 52) | -1.98 (8.10) | -0.42 (6.80) | -0.12 (5.92) | -0.08 (6.73)
  7) Role emotional (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  7) Role emotional (week 26) | -0.54 (7.87) | 0.42 (6.96) | -1.16 (6.60) | -1.01 (6.28)
  7) Role emotional (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  7) Role emotional (week 52) | -1.02 (7.70) | 0.59 (6.89) | -1.05 (8.16) | -1.21 (7.31)
  8) Mental health (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  8) Mental health (week 26) | -1.03 (6.54) | 0.16 (6.66) | -0.41 (7.32) | 0.27 (7.34)
  8) Mental health (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  8) Mental health (week 52) | -1.64 (7.63) | -0.35 (6.68) | 0.27 (7.58) | -0.31 (10.24)
  Physical component summary (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  Physical component summary (week 26) | -0.17 (4.19) | 0.14 (4.27) | -0.23 (5.24) | -0.57 (4.80)
  Physical component summary (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  Physical component summary (week 52) | -0.88 (4.73) | 0.19 (4.91) | -0.03 (5.34) | -0.24 (4.52)
  Mental component summary (week 26): number analyzed (Participants) | 128 | 128 | 128 | 64
  Mental component summary (week 26) | -1.13 (6.54) | -0.07 (5.85) | -0.71 (5.91) | -0.42 (6.04)
  Mental component summary (week 52): number analyzed (Participants) | 127 | 129 | 127 | 63
  Mental component summary (week 52) | -1.52 (7.26) | -0.19 (6.31) | -0.23 (6.15) | -0.74 (8.57)

33. Secondary Outcome: Diabetes Therapy-Related Quality of Life (DTR-QoL): Total Score and Scores for the 4 Domains
Description: DTR-QoL questionnaire is a 29-item patient-reported survey of patient health that measures the influence of diabetes treatment on health related-QoL on 4 domains on individual scale ranges: "Burden on social activities and daily activities", "Anxiety and dissatisfaction with treatment", "Hypoglycemia" and "Satisfaction with treatment" on a 7-point graded response scale. The domain score is calculated from the mean score of the attribute items, and the scoring range is converted to 0 - 100 (best-case response = 100; worst case response = 0). The total score, after simple addition of the item scores, is converted to 0 - 100 (best-case response = 100; worst case response = 0). Change from baseline (week 0) in the scores were evaluated at week 26, week 52. Data based on in-trial observation period is presented. W26 and W52 refer to week 26 and week 52 respectively.
Time Frame: week 0, week 26, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
Number analyzed (Participants) | 131 | 132 | 130 | 65
Score on a scale
  1.Burden on social and daily activities (W26): number analyzed (Participants) | 128 | 128 | 128 | 64
  1.Burden on social and daily activities (W26) | 6.44 (17.59) | 6.93 (18.09) | 4.88 (16.46) | 5.29 (19.65)
  1.Burden on social and daily activities (W52): number analyzed (Participants) | 127 | 129 | 127 | 63
  1.Burden on social and daily activities (W52) | 4.73 (18.69) | 6.81 (18.85) | 5.44 (16.57) | 3.99 (19.25)
  2.Anxiety and dissatisfaction with treatment(W26): number analyzed (Participants) | 128 | 128 | 128 | 64
  2.Anxiety and dissatisfaction with treatment(W26) | 6.54 (18.08) | 10.94 (17.83) | 12.24 (17.41) | 9.24 (20.87)
  2.Anxiety and dissatisfaction with treatment(W52): number analyzed (Participants) | 127 | 129 | 127 | 63
  2.Anxiety and dissatisfaction with treatment(W52) | 0.98 (18.60) | 9.93 (19.61) | 11.37 (18.68) | 3.14 (19.79)
  3.Hypoglycemia (W26): number analyzed (Participants) | 128 | 128 | 128 | 64
  3.Hypoglycemia (W26) | 5.18 (20.62) | 1.95 (18.14) | 2.67 (21.14) | 3.26 (19.82)
  3.Hypoglycemia (W52): number analyzed (Participants) | 127 | 129 | 127 | 63
  3.Hypoglycemia (W52) | 4.20 (19.61) | 1.94 (19.36) | 3.87 (20.70) | -0.66 (23.10)
  4.Satisfaction with treatment(W26): number analyzed (Participants) | 128 | 128 | 128 | 64
  4.Satisfaction with treatment(W26) | 9.67 (19.08) | 10.81 (24.53) | 14.29 (28.11) | 13.15 (24.69)
  4.Satisfaction with treatment(W52): number analyzed (Participants) | 127 | 129 | 127 | 63
  4.Satisfaction with treatment(W52) | 2.46 (19.66) | 7.88 (23.92) | 15.49 (27.01) | 6.35 (26.22)
  Total score(W26): number analyzed (Participants) | 128 | 128 | 128 | 64
  Total score(W26) | 6.74 (13.01) | 7.88 (14.40) | 7.90 (12.72) | 7.18 (15.56)
  Total score(W52): number analyzed (Participants) | 127 | 129 | 127 | 63
  Total score(W52) | 3.31 (13.47) | 7.15 (15.69) | 8.25 (12.81) | 3.44 (14.89)

ADVERSE EVENTS:
Time Frame: Week 0 to week 57 (52 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Dulaglutide 0.75 mg
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/132 | 0/130 | 0/65
Serious Adverse Events (participants affected / at risk) | 9/131 | 4/132 | 7/130 | 1/65
Other Adverse Events (participants affected / at risk) | 65/131 | 79/132 | 84/130 | 36/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=131) | Oral Semaglutide 7 mg (N=132) | Oral Semaglutide 14 mg (N=130) | Dulaglutide 0.75 mg (N=65)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=131) | Oral Semaglutide 7 mg (N=132) | Oral Semaglutide 14 mg (N=130) | Dulaglutide 0.75 mg (N=65)
Abdominal discomfort (Gastrointestinal disorders) | 3 (4) | 6 (8) | 9 (9) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 12 (13) | 16 (16) | 20 (20) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 12 (12) | 6 (6) | 3 (3)
Diabetic retinopathy (Eye disorders) | 6 (6) | 12 (12) | 5 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 10 (10) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 2 (3) | 8 (9) | 0 (0)
Influenza (Infections and infestations) | 9 (9) | 9 (9) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 34 (49) | 39 (63) | 39 (49) | 19 (27)
Nausea (Gastrointestinal disorders) | 7 (8) | 11 (11) | 12 (12) | 6 (9)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (4) | 3 (3) | 5 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT03015220/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT03015220/SAP_001.pdf